CLINICAL TRIAL: NCT03762681
Title: A Randomized, Placebo-controlled,Observer-blinded Study, to Evaluate Safety,Tolerability, Pharmacokinetics and Pharmacodynamics of RO7239958 in Healthy Volunteers and Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study of RO7239958 to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Volunteers and Participants With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to program discontinuation.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP40520; 2018-003530-32 (EudraCT Number)
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose, HV (Experimental): Healthy volunteers will be administered a single dose of RO7239958 or placebo subcutaneously (SC).
  Interventions: Drug: RO7239958; Other: Placebo
- Part 2a: Multi-dose, CHB (Experimental): Participants with chronic hepatitis B will be administered different dose levels of RO7239958 or placebo SC. Dosages will be determined from data collected from Part 1.
  Interventions: Drug: RO7239958; Other: Placebo
- Part 2b: Multi-dose, CHB (Optional) (Experimental): Additional study arm to open based on data collected from Part 2a. Participants with chronic hepatitis B will be administered different doses and frequencies of RO7239958 or placebo SC.
  Interventions: Drug: RO7239958; Other: Placebo

INTERVENTIONS:
Drug: RO7239958 — Solution for injection, subcutaneous use (SC).
Other: Placebo — Sodium chloride solution for injection, SC

SUMMARY:
This study is designed to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple ascending doses in healthy volunteers (HV) and participants diagnosed with chronic hepatitis B (CHB).

ELIGIBILITY:
Inclusion Criteria:

All Parts

-Female participants should be of non-childbearing potential and male participants who are with pregnant partners or partners of childbearing potential must agree to remain abstinent or use contraceptive measures

Part 1 (SAD HV only)

* Healthy, as judged by the Investigator
* Non-smoker (nor tobacco containing products) for at least 90 days prior to dosing on Day 1, and agrees to remain non-smoker during the study

Part 2 (CHB only)

* Positive serum HBsAg status for > 6 months prior to screening
* Serum HBsAg level ≥ 250 IU/mL at screening
* On stable entecavir or tenofovir (alone or in combination) treatment and having received the same drug in the 3 months prior to randomisation
* HBV DNA below the lower limit of quantification (LLQ) for ≥ 6 months prior to screening by local testing, and confirmed at screening
* Screening laboratory values (including hematology, chemistry, urinalysis) within normal ranges
* No past or current diagnosis of cirrhosis

Exclusion Criteria:

All Parts

* History or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological disorders, or diagnosed central or peripheral neurological disease, capable of altering the absorption, metabolism, or elimination of drugs, or constituting a risk when taking the study treatment, or of interfering with the interpretation of the data
* History of lymphoma, leukemia, or malignancy within the past five years
* Positive for human immunodeficiency virus (HIV) infection
* Participant under judicial supervision, guardianship or curatorship

Part 1 (SAD HV only)

* Screening ECG showing clinically relevant abnormalities
* Abnormal blood pressure
* History or presence of liver disease, or known hepatic or biliary abnormalities
* Alanine aminotransferase (ALT) ≥1.5 × upper limit of normal (ULN)
* Any clinically significant out of range findings in other laboratory test results or any other clinically significant (as judged by the Investigator) abnormalities in the physical examination at screening and on Day -1
* Positive for hepatitis B surface antigen (HBsAg), or hepatitis B core total antibody [anti-HBc]), or hepatitis C virus (HCV) antibody test result

Part 2 (CHB only)

* History or presence of bridging fibrosis or cirrhosis or decompensated liver disease
* History or presence of a medical condition associated with liver disease other than HBV infection. Other known hepatic or biliary abnormalities
* History of or suspicion of hepatocellular carcinoma or alpha fetoprotein (AFP) ≥13 ng/mL
* History of having received (in the last six months) or currently receiving any systemic antineoplastic (including radiation) or immune-modulatory treatment (including systemic corticosteroids)
* History of organ transplantation
* Estimated glomerular filtration rate (eGFR) <70 mL/min/1.73m^2
* Confirmed QT interval corrected using Fridericia's formula (QTcF) >450 ms
* Expected to need any other systemic antiviral therapy at any time during participation in the study
* Positive hepatitis C antibody test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Bulgaria (2):
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
  - COMAC Medical; Clinical Research Unit for Phase I, Sofia
- Queen Mary Hospital, Hong Kong, Hong Kong
- Auckland Clinical Studies Limited, Auckland, New Zealand
- ID Clinic, Mysłowice, Poland
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Asan Medical Center., Seoul
- Taiwan (2):
  - Kaohsiung Medical University, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - Royal Liverpool University Hospital, Liverpool
  - King College Hospital NHS Foundation Trust, London
  - Chelsea & Westminster Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Geretti AM, Sostelly A, Buatois S, Lu S, Lemenuel A, Attley G, Bopst M, Alvarez-Sanchez R, Mueller H, Gane E. Safety, pharmacokinetics, and pharmacodynamics of the antisense oligonucleotide RO7239958 in healthy volunteers and adults with chronic hepatitis B infection. Antimicrob Agents Chemother. 2025 Dec 10;69(12):e0067925. doi: 10.1128/aac.00679-25. Epub 2025 Nov 4. PMID 41186228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part 1 all healthy volunteers were enrolled at 1 center in New Zealand. In Part 2a, participants with chronic hepatitis B (CHB) were enrolled at 7 centers across 5 countries: Bulgaria, United Kingdom, Hong Kong, Korea, and New Zealand.
Pre-assignment Details: Part 1, single ascending dose (SAD), enrolled healthy volunteers. In Part 2a, two doses of RO7239958 at two dose levels were administered in participants with CHB. No additional arms were opened in Part 2a. Part 2B of the study was not conducted due to early termination of the study.
Groups:
- Part 1, Cohorts 1-4: Placebo: Healthy volunteers were administered a single dose of placebo subcutaneously (SC).
- Part 1, Cohort 1: 0.1 mg/kg RO7239958: Healthy volunteers were administered a single dose of 0.1 mg/kg RO7239958 SC.
- Part 1, Cohort 2: 0.3 mg/kg RO7239958: Healthy volunteers were administered a single dose of 0.3 mg/kg RO7239958 SC.
- Part 1, Cohort 3: 1.0 mg/kg RO7239958: Healthy volunteers were administered a single dose of 1.0 mg/kg RO7239958 SC.
- Part 1, Cohort 4: 1.5 mg/kg RO7239958: Healthy volunteers were administered a single dose of 1.5 mg/kg RO7239958 SC.
- Part 2a: Placebo: Participants with chronic hepatitis B (CHB) were administered two doses of placebo SC at a dosing frequency of once every four weeks (Q4W).
- Part 2a, Arm 1: 0.2 mg/kg RO7239958: Participants with CHB were administered two doses of 0.2 mg/kg RO7239958 SC at a dosing frequency of Q4W.
- Part 2a, Arm 2: 0.4 mg/kg RO7239958: Participants with CHB were administered two doses of 0.4 mg/kg RO7239958 SC at a dosing frequency of Q4W.
Period: Part 1
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Started | 8 | 8 | 8 | 8 | 8 | 0 | 0 | 0
Completed | 8 | 8 | 8 | 7 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2a
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Started | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pandemic Travel Restrictions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.7) | 36.5 (15.1) | 28.9 (9.1) | 31.8 (14.1) | 28.8 (7.2) | 46.0 (18.4) | 47.5 (7.4) | 45.6 (7.3) | 36.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Male | 7 | 8 | 7 | 8 | 8 | 2 | 8 | 5 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 8 | 7 | 7 | 6 | 8 | 2 | 7 | 5 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 1 | 0 | 0 | 4 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 5 | 7 | 3 | 5 | 6 | 0 | 3 | 4 | 33
  More than one race | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product (including investigational drug) during the course of a clinical investigation. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease that was temporally associated with the use of the investigational product, regardless of whether it was considered to be related to the investigational product or not.
Time Frame: Up to approximately 16 months
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5
Participants | 7 | 3 | 4 | 7 | 5 | 1 | 4 | 1

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs such as systolic and diastolic blood pressure, heart rate, body temperature were evaluated.
Time Frame: Up to approximately 16 months
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Findings
Time Frame: Up to approximately 16 months
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Results
Description: Number of participants with clinically significant abnormalities in clinical laboratory parameters such as serum chemistry, hematology, coagulation, viral serology, urinalysis were evaluated.
Time Frame: Up to approximately 16 months
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5
Participants
  Absolute Neutrophil Count, Low (<10^9/L) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Alanine Transaminase (ALT) or Serum Glutamic Pyruvic Transaminase (SGPT), High | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Aspartate Aminotransferase (AST) or Serum Glutamic-Oxaloacetic Transaminase (SGOT), High | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Injection Site Reactions (ISRs)
Description: Injection site reactions (ISRs) referred to any localized sign or symptom, including pain, erythema, swelling and pruritus and were graded as follows: Grade 1: mild, Grade 2: moderate; Grade 3: severe. Adverse events related to ISRs were reported.
Time Frame: Up to approximately 16 months
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 2 | 8 | 5
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of RO7239958
Time Frame: Part 1: pre-dose on Day 1 and post-dose at 15 minutes (min), 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 30, 36, 48, 72, 96, 120, 168 hours. Part 2a: pre-dose on Days 1 and 29 and post-dose at 30 min, 1, 2, 4, 6, 8, 24 hours.
Population: PK population included all study participants who received active treatment unless there were significant violations of inclusion or exclusion criteria, or if data were unavailable or insufficient to allow for full analysis. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: nanomoles/liter (nmol/L)
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
nanomoles/liter (nmol/L)
  Day 1 | 5.93 (1.37) | 19.9 (5.65) | 102 (43.7) | 166 (64.8) | 9.21 (1.69) | 21.2 (2.96)
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29 |  |  |  |  | 8.81 (3.51) | 19.3 (2.77)

7. Secondary Outcome: Time to Cmax (Tmax) of RO7239958
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
hours (h)
  Day 1 | 1.75 [1.50 to 4.00] | 2.00 [1.53 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.50 to 3.00] | 1.00 [0.50 to 2.00] | 1.00 [1.00 to 2.00]
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29 |  |  |  |  | 2.00 [1.92 to 4.00] | 2.00 [1.00 to 2.00]

8. Secondary Outcome: Area Under the Curve From Time 0 to the Last Measurable Concentration (AUClast) of RO7239958
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
h*nmol/L
  Day 1 | 34.5 (3.07) | 106 (26.4) | 508 (152) | 868 (230) | 59.4 (17.7) | 153 (22.1)
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29 |  |  |  |  | 63.9 (24.6) | 161 (10.1)

9. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC0-24) of RO7239958
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
h*nmol/L
  Day 1 | 33.9 (3.07) | 98.4 (22.6) | 481 (150) | 819 (227) | 54.9 (11.5) | 125 (15.9)
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29 |  |  |  |  | 58.0 (19.9) | 119 (5.36)

10. Secondary Outcome: Half-life (t1/2) of RO7239958
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: h
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
h
  Day 1: number analyzed (Participants) | 8 | 4 | 6 | 5 | 7 | 4
  Day 1 | 5.36 [1.83 to 58.7] | 151 [126 to 293] | 411 [333 to 836] | 515 [305 to 1000] | 3.13 [2.87 to 512] | 499 [395 to 743]
  Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 4
  Day 29 |  |  |  |  | 3.04 [2.67 to 3.87] | 231 [181 to 284]

11. Secondary Outcome: Cumulative Amount of Drug Excreted in Urine (Ae)
Description: The cumulative amount of drug excreted in urine (Ae) over a 24 hour period or over defined time periods linked to the pools of urine collected was analyzed.
Time Frame: Part 1: 0-4 h, 0-8 h, 0-12 h and 0-24 h on Day 1; Part 2a: 0-4 h and 0-8 h on Days 1 and 29
Population: Pharmacokinetic (PK) population included all study participants who received active treatment unless there were significant violations of inclusion or exclusion criteria, or if data were unavailable or insufficient to allow for full analysis. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: micrograms (µg)
Arm/Group | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 5
micrograms (µg)
  Day 1, accumulation interval 0- 4 h | 16.4 (8.87) | 35.4 (33.7) | 104 (72.6) | 290 (272) | 25.0 (14.1) | 81.9 (125)
  Day 1, accumulation interval 0-8 h | 23.1 (12.3) | 50.1 (48.2) | 153 (76.0) | 446 (359) | 35.2 (22.3) | 127 (170)
  Day 1, accumulation interval 0-12 h: number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0
  Day 1, accumulation interval 0-12 h | 23.5 (16.5) | 51.2 (51.0) | 172 (81.3) | 474 (379) |  |
  Day 1, accumulation interval 0-24 h: number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0
  Day 1, accumulation interval 0-24 h | 23.8 (20.0) | 51.7 (55.9) | 189 (92.1) | 497 (383) |  |
  Day 29, accumulation interval 0-4 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29, accumulation interval 0-4 h |  |  |  |  | 23.4 (14.5) | 46.4 (44.4)
  Day 29, accumulation interval 0-8 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 5
  Day 29, accumulation interval 0-8 h |  |  |  |  | 38.1 (23.3) | 85.1 (56.9)

12. Secondary Outcome: Part 2a: Change From Baseline in Hepatitis B Surface Antigen (HBsAg) Levels
Time Frame: Part 2a: Days 1 (pre-dose), 8, 15, 22, 29 (pre-dose); at discontinuation (DC) and at follow-up visits 14, 28, 56, and 84 days after the last dose of study drug (up to 16 weeks)
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: log10[international units (IU)/mL]
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 2 | 8 | 5
log10[international units (IU)/mL]
  Baseline | 3.66 (0.50) | 3.52 (0.61) | 3.22 (0.38)
  Change at Day 8 | -0.20 (0.44) | -0.05 (0.18) | -0.13 (0.16)
  Change at Day 15 | -0.20 (0.27) | -0.05 (0.31) | -0.13 (0.17)
  Change at Day 22 | -0.40 (0.40) | -0.05 (0.12) | -0.17 (0.23)
  Change at Day 29 | -0.06 (0.19) | -0.09 (0.11) | -0.08 (0.23)
  Change at Day 43 | 0.04 (0.02) | -0.11 (0.35) | -0.26 (0.33)
  Change at Day 57 | 0.05 (0.01) | -0.12 (0.30) | -0.19 (0.26)
  Change at Day 85: number analyzed (Participants) | 2 | 8 | 4
  Change at Day 85 | -0.01 (0.09) | -0.14 (0.24) | -0.06 (0.08)
  Change at Day 113: number analyzed (Participants) | 1 | 7 | 4
  Change at Day 113 | 0.23 (NA) — SD was not estimable for 1 participant. | -0.03 (0.09) | -0.05 (0.09)

13. Secondary Outcome: Part 2a: Change From Baseline in Hepatitis B Surface Antibody (Anti-HBs) Levels
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: log10[IU/mL]
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 2 | 8 | 5
log10[IU/mL]
  Baseline | 0.48 (0.00) | 0.50 (0.08) | 0.48 (0.00)
  Change at Day 8 | 0.00 (0.00) | 0.02 (0.05) | 0.00 (0.00)
  Change at Day 15 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Day 22 | 0.00 (0.00) | 0.02 (0.06) | 0.00 (0.00)
  Change at Day 29 | 0.00 (0.00) | 0.01 (0.04) | 0.00 (0.00)
  Change at Day 43 | 0.00 (0.00) | 0.02 (0.05) | 0.00 (0.00)
  Change at Day 57 | 0.00 (0.00) | 0.02 (0.06) | 0.00 (0.00)
  Change at Day 85: number analyzed (Participants) | 2 | 8 | 3
  Change at Day 85 | 0.00 (0.00) | 0.02 (0.07) | 0.00 (0.00)
  Change at Day 113: number analyzed (Participants) | 1 | 7 | 4
  Change at Day 113 | 0.00 (NA) — SD was not estimable for 1 participant. | 0.02 (0.06) | 0.00 (0.00)

14. Secondary Outcome: Part 2a: Number of Participants With HBsAg Loss
Description: HBsAg loss was defined as a measurement below the lower limit of sensitivity.
Time Frame: as for outcome 12
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 2 | 8 | 5
Participants | 0 | 0 | 0

15. Secondary Outcome: Part 2a: Number of Participants With Hepatitis B Envelope Antigen (HBeAg) Loss in HBeAg-positive Participants
Description: HBeAg loss was defined as a measurement below lower limit of sensitivity. Positive HBeAg is a marker of an actively replicating HBV virus infection.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 0 | 3 | 0
Participants
  HBeAg Loss at Baseline |  | 0 |
  HBeAg Loss at Day 8 |  | 0 |
  HBeAg Loss at Day 15 |  | 0 |
  HBeAg Loss at Day 22 |  | 0 |
  HBeAg Loss at Day 29 |  | 0 |
  HBeAg Loss at Day 43 |  | 0 |
  HBeAg Loss at Day 57 |  | 0 |
  HBeAg Loss at Day 85 |  | 0 |
  HBeAg Loss at Day 113 |  | 0 |

16. Secondary Outcome: Part 2a: Number of Participants With Hepatitis B e Antibody (Anti-HBe) Seroconversion in HBeAg-positive Participants
Description: Anti-HbBe was defined as an antibody to HBeAg. Positive HBeAg is a marker of an actively replicating HBV virus infection.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 0 | 3 | 0
Participants
  Anti-HBe Seroconversion at Baseline |  | 0 |
  Anti-HBe Seroconversion at Day 8 |  | 0 |
  Anti-HBe Seroconversion at Day 15 |  | 0 |
  Anti-HBe Seroconversion at Day 22 |  | 0 |
  Anti-HBe Seroconversion at Day 29 |  | 0 |
  Anti-HBe Seroconversion at Day 43 |  | 0 |
  Anti-HBe Seroconversion at Day 57 |  | 0 |
  Anti-HBe Seroconversion at Day 85 |  | 0 |
  Anti-HBe Seroconversion at Day 113 |  | 0 |

17. Secondary Outcome: Part 2a: Number of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Below the Assay Lower Limit of Quantification
Description: Participants with HBV DNA below the assay lower limit of quantification i.e. LLOQ <20 IU/ml at each time-point were analyzed.
Time Frame: Part 2a: Day 1 (pre-dose), 15, 29 (pre-dose); at discontinuation (DC), rebound and at follow-up visits 14, 28, 56, and 84 days after the last dose of study drug (up to 16 weeks)
Population: Safety population included all study participants who received at least one dose of RO7239958 or placebo. Data are reported for participants HBeAg positive or negative at baseline. Number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: participants
Arm/Group | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
Number analyzed (Participants) | 2 | 8 | 5
participants
  HBeAg+: Baseline: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Baseline |  | 3 |
  HBeAg-: Baseline: number analyzed (Participants) | 2 | 5 | 5
  HBeAg-: Baseline | 2 | 5 | 5
  HBeAg+: Day 15: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Day 15 |  | 3 |
  HBeAg-: Day 15: number analyzed (Participants) | 2 | 5 | 5
  HBeAg-: Day 15 | 2 | 4 | 5
  HBeAg+: Day 29: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Day 29 |  | 3 |
  HBeAg-: Day 29: number analyzed (Participants) | 2 | 5 | 5
  HBeAg-: Day 29 | 2 | 5 | 5
  HBeAg+: Day 43: number analyzed (Participants) | 0 | 2 | 0
  HBeAg+: Day 43 |  | 2 |
  HBeAg-: Day 43: number analyzed (Participants) | 2 | 5 | 5
  HBeAg-: Day 43 | 2 | 5 | 5
  HBeAg+: Day 57: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Day 57 |  | 3 |
  HBeAg-: Day 57: number analyzed (Participants) | 2 | 5 | 4
  HBeAg-: Day 57 | 2 | 5 | 4
  HBeAg+: Day 85: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Day 85 |  | 3 |
  HBeAg-: Day 85: number analyzed (Participants) | 2 | 5 | 4
  HBeAg-: Day 85 | 2 | 5 | 4
  HBeAg+: Day 113: number analyzed (Participants) | 0 | 3 | 0
  HBeAg+: Day 113 |  | 3 |
  HBeAg-: Day 113: number analyzed (Participants) | 1 | 4 | 4
  HBeAg-: Day 113 | 1 | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Description: Safety population included all study participants who received at least one dose of RO7239958 or placebo.
Arm/Group | Part 1, Cohorts 1-4: Placebo | Part 1, Cohort 1: 0.1 mg/kg RO7239958 | Part 1, Cohort 2: 0.3 mg/kg RO7239958 | Part 1, Cohort 3: 1.0 mg/kg RO7239958 | Part 1, Cohort 4: 1.5 mg/kg RO7239958 | Part 2a: Placebo | Part 2a, Arm 1: 0.2 mg/kg RO7239958 | Part 2a, Arm 2: 0.4 mg/kg RO7239958
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/2 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/2 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 7/8 | 3/8 | 4/8 | 7/8 | 5/8 | 1/2 | 4/8 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Cohorts 1-4: Placebo (N=8) | Part 1, Cohort 1: 0.1 mg/kg RO7239958 (N=8) | Part 1, Cohort 2: 0.3 mg/kg RO7239958 (N=8) | Part 1, Cohort 3: 1.0 mg/kg RO7239958 (N=8) | Part 1, Cohort 4: 1.5 mg/kg RO7239958 (N=8) | Part 2a: Placebo (N=2) | Part 2a, Arm 1: 0.2 mg/kg RO7239958 (N=8) | Part 2a, Arm 2: 0.4 mg/kg RO7239958 (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT03762681/Prot_SAP_000.pdf